CLINICAL TRIAL: NCT06167525
Title: Assessment of the Effects of Maladaptive Neck Posturing in Surgeons During Microsurgery Procedures Using Upright Go 2 Device
Brief Title: Neck Posturing in Surgeons During Microsurgery Procedures Using Upright Go 2 Device
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Royal College of Surgeons, Ireland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RCSI sponsorship ref: 23-161
Record Dates: First submitted 2023-11-15; First posted 2023-12-12 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Neck Pain Musculoskeletal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neck posture monitoring device without feedback option (Other): Real-time feedback through the device. For surgeons who consent, bio-feedback signals will be given once deviated from a neutral posture for >1 minute.
  Interventions: Device: Real-time feedback through the device. Bio-feedback signals will be given once deviated from a neutral posture for >1 minute. Response of surgeons to bio-feedback signals will be recorded

INTERVENTIONS:
Device: Real-time feedback through the device. Bio-feedback signals will be given once deviated from a neutral posture for >1 minute. Response of surgeons to bio-feedback signals will be recorded — During the first stage of the study the device will be set to record cervical spine positioning without bio-feedback signals. This will be used to record duration of time surgeons held maladaptation postures.
  The second stage will involve real-time feedback through the device. For surgeons who consent, bio-feedback signals will be given once deviated from a neutral posture for >1 minute. Response of surgeons to bio-feedback signals will also be recorded.
  The Neck Disability index score will be used to assess for neck pain and the functional implications in relation to reported neck pain. This will be completed following study completion.

SUMMARY:
Consultant and senior registrars performing microsurgery will be invited to participate in this Study. The study will take place at single site (Beaumont Hospital). A questionnaire to collect demographic information (age, height, sex, year of training, prior neck trauma or know neck issues) will be given to the consented surgeons. Additionally, surgery characteristics will be recorded (procedure, surgeon role (i.e lead or assisting), table height, frequency of adjustment of table height, and use of sitting or step stool, headlight, and/or loupes for >50% of the procedure).

A postural training device, Upright Go 2 will be positioned at the spinous process of the cervical vertebrae of each surgeon and used to measure neck positions during microsurgical procedures. The device will be calibrated to an ideal neutral cervical spine position, so that excessive flexion and extension of the neck can be recorded.

The device contains built-in sensors that provide bio-feedback in the form of gentle vibrations if posture has deviated from neutral position.

During the first stage of the study the device will be set to record cervical spine positioning without bio-feedback signals. This will be used to record duration of time surgeons held maladaptation postures.

The second stage will involve real-time feedback through the device. For surgeons who consent, bio-feedback signals will be given once deviated from a neutral posture for >1 minute. Response of surgeons to bio-feedback signals will also be recorded.

The Neck Disability index score will be used to assess for neck pain and the functional implications in relation to reported neck pain. This will be completed following study completion.

ELIGIBILITY:
Inclusion Criteria:

* Plastic and reconstructive surgeons performing microsurgery
* Consultants, Registrars, and Senior House Officers with no prior cervical spine surgery or cervical degeneration

Exclusion Criteria:

* Surgeons not performing microsurgery on a regular basis (at least once a month)
* Plastic and reconstructive surgery trainees with <1 years experience in microsurgery.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-01-18 (Estimated); Primary Completion 2024-04-10 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Measuring neck positioning using upright go 2 device during microsurgery procedures and adjustments in neck positioning after receiving bio-feedback signals. | 3 months
  1. The Upright go 2 device has sensors that are used to detect neck posture in real-time. This device will be used to measure surgeon's postural maladaptation. This measure will be degree angle of cervical spine flexion (>30 degrees is considered maladaptive)
  2. Neck Disability Index to assess neck pain and condition-specific functional status which will be compared to neck posture data obtained from neck measuring device. Score of 10-28% (i.e., 5-14 points) is considered by the authors to constitute mild disability; 30-48% is moderate; 50-68% is severe; 72% or more is complete.
  Measure of change will be baseline (i.e no bio-feeback) and bio-feeback through device. Time between baseline and bio-feedback will depend on when each participant has a microsurgical case.
Time and rate spent in maladaptive neck positions in surgeons during as measured by the upright go 2 device. | 3 months
  1. Feedback from device will be recorded (amount of times feedback is required and whether surgeons react to biofeedback). Again measure in degree angles of cervical flexion and adjustment angle.
  This information will indicate the amount of times adjustments are made in neck positioning by the participants and if responses to bio-feeback are continuous and sustained.

IPD SHARING:
Plan to Share IPD: No
Study aims have been described so that data relevant to the aims of the study is collected by researchers. Data for all questionnaires will be stored in numerical value without context to their significance in the database.
  Paper versions of the questionnaires will be used to collect the scores during in-person meeting with one of the project investigators. These paper sheets will be discarded in the hospital confidentiality bins in Beaumont Outpatients after the data is transferred to the database